CLINICAL TRIAL: NCT04447937
Title: Analysis of Medical Therapy and History as Risks of Immunodeficiency in Multiple Sclerosis Patients
Brief Title: Immunodeficiency in MS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Advanced Neurosciences Institute (Other)
Collaborators: Novel Pharmaceutics Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: NPI-110
Record Dates: First submitted 2020-06-12; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Multiple Sclerosis; Hypogammaglobulinemia; Immunodeficiency; Infection, Bacterial
MeSH Terms: conditions — Multiple Sclerosis; Agammaglobulinemia; Immunologic Deficiency Syndromes; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Sclerosis and Related Diseases: Individuals with one or more immunoglobulin level results and medical histories available for data collection will be included. Subjects will be 18 years of age or older at the time of data collection.
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — There are no interventions associated with the study.

SUMMARY:
The purpose of this study is to identify if there is a relationship between multiple sclerosis disease-modifying therapy exposure, immunodeficiencies, and infection risk in subjects living with MS.

DETAILED DESCRIPTION:
The purpose of this study is to identify if there is a relationship between multiple sclerosis disease-modifying therapy exposure, immunodeficiencies, and infection risk in subjects living with MS. By understanding this relationship future studies can be designed to create a model of immunosenescence in multiple sclerosis, which could help healthcare providers to predict and assess health risks. Preventative strategies can then be tested to look for ways to prevent these immune-related risks.

ELIGIBILITY:
Inclusion Criteria

* One or more immunoglobulin level results and medical history available
* 18 years of age or older at the time of data collection
* Patients with first symptom MS or other isolated demyelinating syndromes, neuromyelitis optica, or rheumatic-associated CNS inflammation

Exclusion Criteria:

* No evidence of CNS autoimmune disease
* Less than 18 years of age at the time of data abstraction
* Undergoing plasma exchange at the time of any lab tests drawn

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective data from 1500 patients with immune-mediated CNS disease is expected to be used from the electronic medical record eClinicalWorks and other electronic and paper archives of Advanced Neurosciences Institute.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-06-29 (Estimated); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Immunoglobulin Levels | 1 year
  IgG, IgA, IgM

SECONDARY OUTCOMES:
Infections | 1 year
  Serious and non-serious
Immune-mediated conditions | 1 year
  Serious and non-serious
Malignant and pre-malignant conditions | 1 year
  Serious and non-serious

CONTACTS AND LOCATIONS:
Overall Officials: Samuel F Hunter, MD, PhD, Principal Investigator — Advanced Neurosciences Institute
Locations (1):
- Advanced Neurosciences Institute, Franklin, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Publications and findings from research